CLINICAL TRIAL: NCT01337466
Title: Biodistribution and Dosimetry of [124i]FIAU in Patients With Prosthetic Joint Infection of The Knee or Hip and Healthy Subjects Using PET-CT Scanning
Brief Title: Biodistribution and Dosimetry Evaluation of [124I]FIAU
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioMed Valley Discoveries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BVD001
Record Dates: First submitted 2011-04-08; First posted 2011-04-19 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Prosthesis Related Infections
Keywords: Phase I; FIAU; Fialuridine; Biodistribution; Dosimetry; Prosthetic; Joint; Infection; PET-CT
MeSH Terms: conditions — Prosthesis-Related Infections; Infections | interventions — fialuridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [124I]FIAU (Experimental): single dose study of [124I]FIAU in healthy volunteers or subjects with prosthetic joint infection who will undergo PET-CT scanning
  Interventions: Radiation: [124I]FIAU

INTERVENTIONS:
Radiation: [124I]FIAU — This is a single dose study of 2 mCi [124I]FIAU in healthy volunteers or subjects with prosthetic joint infection of the knee or hip who will undergo serial PET-CT scanning.
  Other Names: Fialuridine

SUMMARY:
This protocol will evaluate the biodistribution and dosimetry of [124I]FIAU in both healthy volunteers and patients with prosthetic joint infections. This pilot study will also investigate the safety and tolerability of [124I]FIAU.

ELIGIBILITY:
The following are the main inclusion criteria for all subjects:

1. Males or females age > 18 years
2. Informed consent
3. Subjects with chronic medical conditions such as hypertension and diabetes should be considered stable by the principal investigator
4. Women should be postmenopausal or surgically sterile
5. Able to return for all study assessments

In addition, the following main inclusion criteria apply for subjects with suspected prosthetic joint infection:

1. Operative intervention planned in the 30 days following study enrollment
2. Prosthetic joint implant in site for more than 3 months prior to enrollment

The following are the main exclusion criteria for all subjects:

1. Unable to comply with study requirements
2. Indication in the opinion of the principal investigator for surgery within 48 hours of presentation.
3. Receipt of any antibiotic therapy in the 2 weeks preceding imaging
4. Immunosuppression, e.g., human immunodeficiency virus (HIV) infection, s/p organ transplantation, receipt of steroids for > 10 days at > 10 mg of prednisone equivalent daily within the 90 days prior to enrollment
5. Requirement for any medication that predisposes to lactic acidosis (e.g., metformin, iron, isoniazid and salicylates; see Appendix A)
6. Requirement for any medication that has potential mitochondrial toxicity, e.g., nucleoside analogues (zidovudine, didanosine, stavudine)
7. History of an inherited mitochondrial disorder (e.g., Leber's hereditary neuropathy, neuropathy, ataxia, retinitis pigmentosa and ptosis [NARP], myoneurogenic gastrointestinal encephalopathy [MNGIE], myoclonic epilepsy with ragged red fibers [MERFF] and mitochondrial myopathy, encephalomyopathy, lactic acidosis and stroke-like syndrome [MELAS]
8. Chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
9. Pre-existing myopathy or neuropathy
10. Abnormal liver function tests defined as alanine aminotransferase (ALT) > the upper limit of normal (ULN), aspartate aminotransferase (AST) > ULN, gamma glutamyl transferase (GGT) > ULN
11. Alcohol use > 3 units per day in men or 2 units per day in women or active intravenous drug use
12. Creatinine clearance < 30 mL/min
13. Body mass index > 40
14. Life expectancy < 6 months
15. Hypersensitivity to iodine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Determine the biodistribution and dosimetry evaluation of [124I]FIAU | 72 hrs
  Subjects will be dosed with [124I]FIAU at Time 0 on Day 0, and a PET-CT scan will be conducted immediately after the injection. Imaging will be repeated at 2 hours, 4 hours, 6 hours, 24 hours, 48 hours, and 72 hours after dosing.
  All images generated will be reviewed for biodistribution and dosimetry.

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of [124I]FIAU | 28 +/- 2 days
  Safety will be monitored throughout the study for all subjects. Safety will be assessed by monitoring of adverse events and vital signs, clinical laboratory tests including LFTs, lactate, serum chemistry and CBC, physical examination, and 12-lead ECG.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Mont, MD, Principal Investigator — Sinai Hospital of Baltimore
Locations (3):
- United States (3):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - North Shore long Island Jewish Medical Center, Lake Success, New York